CLINICAL TRIAL: NCT05699694
Title: Open-labeled Pilot Study on the Efficacy of a New Food Supplement Composed of Natural Stem Cell Mobilizers for the Improvement of Motor Performance and Quality of Life in Parkinsonian Patients
Brief Title: Clinical Study on the Efficacy of Natural Stem Cell Mobilizers on Parkinson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sociedad Española de Medicina Regenerativa y Terapia Celular (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13246
Record Dates: First submitted 2023-01-11; First posted 2023-01-26 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Stemregen (Experimental): Experimental product encapsulated will be consumed orally with a glass of water. Six capsules per day will be consumed daily for 6 months.
  Interventions: Dietary Supplement: StemRegen product

INTERVENTIONS:
Dietary Supplement: StemRegen product — Products will be consumed orally in capsules with a glass of water. Six capsules per day will be consumed daily for 6 month. Two main administration schedules are possible:
  Two in the morning, 2 at noon, and 2 in the evening at each meal depending on individual habits of the volunteers to reduce non-compliance.

SUMMARY:
Parkinson's disease is defined as the progressive loss or deterioration of dopaminergic neurons, Treatment approaches to maintain the normal dopamine level that include medication, surgery, cell therapy supplementation of L-Dihydroxyphenylalanine (L-Dopa), a precursor of dopamina, Stem cells from bone marrow can be mobilized according to the need of repair of the tissue. Suggested use of the food supplement actually sold in the USA and in Europe: Take two capsules, 1 to 3 times per day with a glass of water. Increase the Stem Cell circulating in the peripheral blood.

DETAILED DESCRIPTION:
Parkinson's disease is defined as the progressive loss or deterioration of dopaminergic neurons in Substantia Nigra (SN) of the brain. These cells normally produce dopamine which acts like a messenger for normal muscular movement. Having less quantity of dopamine in the synaptic cleft due to the loss of neural cells, symptoms become apparent. Neuroinflammation and oxidative stress are involved. Treatment approaches to maintain the normal dopamine level that include medication, surgery, cell therapy supplementation of L-Dihydroxyphenylalanine (L-Dopa), a precursor of dopamine, in the form of Levodopa and/or Carbidopa, has been available for PD therapy for 50 years. Stem cells constitute the repair system of the body. Stem cells from bone marrow can be mobilized according to the need of repair of the tissue. Suggested use of the food supplement actually sold in the USA and Europe: Take two capsules, 1 to 3 times per day with a glass of water.

All raw materials are food grade. All extracts are water or ethanolic extracts, which are authorized solvents for dietary supplements in the USA and EU. All ingredients are compliant with US and EU contaminants regulation (microbiological profile, heavy metals, pesticides) especially EU pharmacopeia, the product shows to increase Stem Cell circulation in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Adults from both genders
* Diagnosed by neurologist or qualified health care practitioner with PD for 5 years or more
* Stabilized symptomatic treatment for PD for more than 3 months
* Age: over 21 years old
* Volunteers able to understand the nature of the study and to sign a written consent form

Exclusion Criteria:

* Gastro-intestinal surgery that may modify or decrease the intestinal absorption of nutrient and experimental product
* Serious traumatism in the last 3 months
* Heavy surgery operation in the last 3 months
* Non-controlled evolutive disease
* Drug or medication abuse in the last 2 years
* History of non-compliance in previous studies
* Regular consumption of similar ingredients or food supplements compared to experimental product in the past 3 months
* Any medical problem or trouble identified by the investigator that could alter the capacity of the volunteer to end the study
* Any drug medication that could mask, decrease or interfere experimental product efficacy
* Surgery operation planned during the year
* Breastfeeding, pregnant women
* Known allergies to one of the ingredients entering in the composition of the experimental product
* Severe liver and renal failure
* Actual participation to another clinical trial

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 6 months
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Parkinson's Disease (PD) symptoms: Change from Baseline | 6 months
  UPDRS questionnaire which represents a validated and standardized questionnaire for PD diagnostic and disease progression evaluation: 0=normal - 4= Severe
Quality of Life Assessed by the Parkinson's Disease | 6 Months
  Modified SF-36 quality of life assessment from Dr Gitte Jensen used in several clinical studies at NIS labs clinical center, Oregon USA, result from excellent to Terrible
Parkinson's Disease (PD) symptoms: Change | 6 months
  Schwab and England activities of daily living activities scales from 0% to 100%

CONTACTS AND LOCATIONS:
Overall Officials: Miguel G Garber, MD, Principal Investigator — Healthy Longevity Clinic; Felix Pedrero Ramallo, MD, Study Chair — Clinica Castello 68; Christian Drapeou, PhD, Study Director — Kalyagen
Locations (1):
- Clinica Castello 68, Madrid, Spain